CLINICAL TRIAL: NCT05177133
Title: Anti-PD-1, Capecitabine, and Oxaliplatin for the First-line Treatment of dMMR Esophagogastric Cancer (AuspiCiOus-dMMR): a Proof-of-principle Study
Brief Title: Anti-PD-1 and CapOx for the First-line Treatment of dMMR Esophagogastric Cancer (AuspiCiOus)
Acronym: AuspiCiOus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Hanneke W. M. van Laarhoven, prof. dr. H.W.M. van Laarhoven, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL77094.018.21
Record Dates: First submitted 2021-09-07; First posted 2022-01-04 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Gastric Adenocarcinoma; Esophageal Adenocarcinoma
Keywords: Advanced esophagogastric cancer; Infiltrating immune cells; IFNy expression; chemotherapy; immunotherapy; Microsatellite instability
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Microsatellite Instability | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Capecitabine, oxaliplatin and retifanlimab (Experimental): IV and PO Capecitabine 1000 mg/m2, oxaliplatin 130 mg/m2, every three weeks (up to 2 cycles) IV retifanlimab 500mg, every four weeks
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Retifanlimab

INTERVENTIONS:
Drug: Capecitabine — PO Capecitabine
  Other Names: Xeloda
Drug: Oxaliplatin — IV Oxaliplatin
  Other Names: Oxaliplatin Accord
Drug: Retifanlimab — IV retifanlimab
  Other Names: INCMGA00012

SUMMARY:
To investigate the effects of the combination of two chemotherapies followed by immunostimulants on the interferon gamma expression and infiltration of cytotoxic T cells in the tumour microenvironment in patients with previously untreated metastatic or locally advanced esophagogastric cancer.

DETAILED DESCRIPTION:
This is a multi-center, open label, proof-of-principle study for patients with previously untreated metastatic or locally advanced esophagogastric cancer. Patients are sequentially treated with standard of care capecitabine and oxaliplatin, and retifanlimab. Patients are treated with 2 cycles of CapOx (1 cycle is 3 weeks) and sequentially with 4-weekly cycles of retifanlimab up to 2 years. The investigators will include 25 patients in this study.

Biopsies, blood and faeces will be collected during treatment for assessment of infiltrating immune cells and IFNy expression, as well as for other translational research purposes. CT scans are made for evaluation of tumor response before and after chemotherapy, and after 2-3 cycles of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent according to ICH/GCP, and national/local regulations prior to any screening procedures.
* Male or female adult patients (≥ 18 years).
* Patients with histologically confirmed diagnosis of metastatic or irresectable HER2 negative adenocarcinoma of the stomach or gastroesophageal junction (Siewert II and III); patients with HER2 positive disease are eligible when treatment with trastuzumab is contraindicated. If histology cannot be obtained, cytology is acceptable to prove metastatic disease.
* Patients with metastatic or irresectable adenocarcinoma of the stomach or oesophagus not pre-treated with chemotherapy or radiotherapy for irresectable or metastatic disease. Palliative radiotherapy on the primary tumor or a metastatic lesion is allowed if other untreated lesions eligible for evaluation are present.
* Measurable disease as assessed by RECIST 1.1
* dMMR identified by IHC of mismatch repair proteins MLH1, PMS2, MSH2 en MSH6
* Primary tumor or metastasis accessible for repeat fresh histological biopsies
* ECOG (WHO) performance status 0-2
* Patient has adequate bone marrow and organ function as defined by the following laboratory values:

  * Absolute Neutrophil Count (ANC) > 1.5 x 109 /L
  * Hemoglobin (Hgb) > 5.6 mmol/L
  * Platelets > 100 x 109 /L
* Serum total bilirubin within ≤ 1.5 x ULN (upper limit of normal); or total bilirubin < 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert's syndrome; biliary drainage is allowed for biliary obstruction
* Serum creatinine < 1.5 x ULN or creatinine clearance >30 mL/min/1.73 m2
* Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) < 2.5x ULN within normal range or < 5.0 x ULN if liver metastases are present
* If a female patient is of child-bearing potential, as evidenced by regular menstrual periods, she must have a negative pregnancy test (urine or serum; beta-human chorionic gonadotropin (β-hCG)) documented prior to the first administration of study drug. If sexually active, the patient must agree to use contraception considered adequate and appropriate by the Investigator during the period of administration of study drug and after the end of treatment as recommended.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Exclusion Criteria:

* Severe renal impairment (CLcr ≤ 30 ml/min)
* Any clinically significant disorder impacting the risk-benefit balance negatively per physician's judgment.
* Any prior anti-cancer chemotherapy, biologic or investigational therapy for metastatic or irresectable stomach or oesophageal cancer
* Disease progression within six months after completion of (neo)adjuvant chemotherapy containing a fluoropyrimidine and/or platinum compound. (Disease progression within 6 months after completion of neoadjuvant chemoradiation carboplatin AUC 2 and paclitaxel 50 mg/m2 is allowed.)
* All target lesions in a radiation field without documented disease progression.
* Patient has known brain metastases, unless previously treated and well-controlled for at least 3 months (defined as clinically stable, no edema, no steroids and stable in 2 scans at least 4 weeks apart).
* Past or current malignancy other than entry diagnosis interfering with prognosis of metastatic gastroesophageal cancer.
* Known uncontrollable hypersensitivity or contraindications to any of the components of retifanlimab, fluoropyrimidines, leucovorin, oxaliplatin. Patients with previous dose reductions or delays are eligible.
* Complete dihydropyrimidine dehydrogenase deficiency.
* Patient has active, uncontrolled bacterial, viral or fungal infection(s) requiring systemic therapy.
* Patient has known past or active infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
* Signs of interstitial lung disease (ILD)
* Participants with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment contraindicate patient participation in the clinical study.
* Use of other investigational drugs within 30 days of enrollment.
* Patient is enrolled in any other clinical protocol or investigational trial that will interfere with the primary endpoint of the current study.
* Patients who in the investigators' opinion may be unwilling, unable or unlikely to comply with requirements of the study protocol.
* Breast feeding, known pregnancy, positive serum pregnancy test or unwillingness to use a reliable method of birth control, during therapy and for 3 months following the last dose of study treatment.
* Treatment within 4 weeks with DPD inhibitors, including sorivudine or its chemically related analogues such as brivudine.
* Pre-existing motor or sensory neurotoxicity greater than CTCAE grade 1.
* History of organ transplant, including allogeneic stem cell transplantation.
* Receiving probiotics as of the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2029-11-04 (Estimated)

PRIMARY OUTCOMES:
Effect of chemo- and immunotherapy on the interferon gamma expression signature in the tumor microenviornment | 40 months
  RNA expression analysis (Nanostring) to determine changes in Interferon gamma expression signature before and during treatment
Effect of chemo- and immunotherapy on the immune infiltrate in the tumor microenvironment | 40 months
  Flow cytometry to determine changes in immune infiltrate in the tumor before and during treatment
Effect of chemo- and immunotherapy on the immune infiltrate on the tumor microenvironment | 40 months
  Multicolor immunohistochemstry to determine changes in immune infiltrate in the tumor before and during treatment

SECONDARY OUTCOMES:
Overall survival | 60 months
  Determine overall survival of patients within the study
Overall survival | 60 months
  Compare overall survival with a propensity score matched cohort
Progression free survival (PFS) | 60 months
  Assess the PFS of patients within the study
Progression free survival (PFS) | 60 months
  Compare PFS with a propensity score matched cohort
Response rate | 60 months
  Determine response rate by comparing RECIST evaluation of CT scans before and during treatment
Adverse events | 60 months
  To determine adverse events of CapOx and retifanlimab
Measure PROMs via established PROFILES | 60 months
  Patient reported outcome measures (PROMs) are measured with the established PROFILES infrastructure (Patient Reported Outcomes Following Initial treatment and Long term Evaluation of Survivorship). PROMs will be assessed and compared at baseline and throughout treatment
Percentage subsequent treatment lines | 60 months
  The percentage of patients proceeding to subsequent lines of treatment after progression

OTHER OUTCOMES:
Impact of cytotoxic therapy and PD-1 inhibition on the anti-tumor immune respons | 40 months
  Assess changes in RNA expression (Nanostring) in peripheral blood mononuclear cells (PBMCs) before and during treatment
Impact of cytotoxic therapy and PD-1 inhibition on the anti-tumor immune respons | 40 months
  Percentage tumor and immune cells in tumor tissue
Phenotype of PBMCs | 40 months
  Determine change in phenotype of PBMCs with flow cytometry, before and after chemotherapy
Immunohistochemistry | 40 months
  Perform immunohistochemistry on tumor tissue to determine relative increase of infiltrating immune cells
Stromal markers in tumor | 40 months
  Assess changes in expression level of ADAM12 in tumor tissue
ctDNA | 40 months
  Assess changes in concentration of circulating tumor (ct)DNA in blood
Fecal microbiome | 40 months
  Change in composition of the fecal microbiome by DNA sequencing as a potential biomarker for response to treatment
Cytokine and chemokine release profile | 40 months
  Assess changes in cytokine and chemokine profile in blood with Luminex bead fluorescence assay before and during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jan M Prins, MD, PhD, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Hanneke WM van Laarhoven, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Sarah Derks, Principal Investigator — VU Medisch Centrum - Vrije Universiteit
Locations (8):
- Netherlands (8):
  - Academic Medical Center, Medical Oncology, Amsterdam
  - Amsterdam UMC, location VUmc, Amsterdam
  - Catharina ziekenhuis, Eindhoven
  - Medisch Centrum Leeuwarden, Leeuwarden
  - LUMC, Leiden
  - Radboud UMC, Nijmegen
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht